CLINICAL TRIAL: NCT04061967
Title: Research Project on Reminders and Self-Sampling Can Increase Participation in Gynecology Cell Sampling - Preventive Examination Against Cervical Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, Miriam Elfström, Affiliated Researcher, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-03166
Record Dates: First submitted 2019-08-18; First posted 2019-08-20 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Cervical Cancer; Uterine Cervical Neoplasm; Uterine Neoplasms; Genital Neoplasm; Genital Neoplasm, Female; Uterine Diseases; Genital Diseases, Female; Neoplasms by Site; Neoplasms; Uterine Cervical Disease
Keywords: participation; self sampling; screening
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Neoplasms; Genital Neoplasms, Female; Uterine Diseases; Genital Diseases, Female; Neoplasms by Site; Neoplasms; Uterine Cervical Diseases

STUDY DESIGN:
Intervention Model Description: Adaptive trial that improves the method for improving attendance each year. The first three years of intervention (2019-2021) have been evaluated and is published (Arroyo Mühr, L.S., Wang, J., Hassan, S.S., et al. Int J Cancer. 156. 379-388. 2025). Trial continues with annual enrollment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HPV self sampling test ordered (Other): An invitation to order a HPV self sampling test through an online application will be sent by SMS or electronic letter.
  Interventions: Other: Sending of screening summon.

INTERVENTIONS:
Other: Sending of screening summon. — 2019-2021 - A Cobas PCR Female swab sample packet will be sent. Response rates (participation) will be measured.
  2022 and onwards - A FLOQSwab and corresponding sample tube for analysis on the BD COR platform will be sent.
  Other Names: Response to screening summon.

SUMMARY:
Prevention of cervical cancer with cervical screening is one of the most successful screening activities in medicine. In Sweden, screening was implemented in the 1960s and has since prevented tens of thousands of women from having cervical cancer. Individual invitations to screening result in increased attendance therefore evaluating strategies for reaching women through invitations is particularly valuable. Women who regularly attend screening following an invitation reduce their risk of cervical cancer by as much as 90%. Of the women who are diagnosed with cervical cancer (about 550 women per year in Sweden), as many as 38% did not participate in the screening. Invitations for screening are sent to the entire population in Sweden aged 23-70. The current coverage of screening is 82.9%, which represents the proportion of women ages 23-70 who attend according to recommendations. In addition, many women are sporadic attenders who reduce their risk for cancer somewhat. The highest cancer risk is seen among those women who have never participated as well as women who have had a history of precancerous lesions or HPV infection but have not been followed-up. Cervical cancer is the first form of cancer for which there are approved molecular screening tests (HPV test). Unlike the older screening method (cytology), self-collected samples can be analyzed for HPV (the analysis method is so sensitive that it does not matter if the sample is not optimally taken).

Invitations and reminders about cervical screening are sent by letter to the woman's home address (about 3 million letters per year in Sweden). This strategy results in a waste of resources and has a negative environmental impact. Regarding reminders, we have seen in previous research that the effect is not optimal. When sending a physical reminder letter to women who have not participated in more than 10 years (current routine), only 2% of the women invited came for sampling. Reminders with SMS are now standard for many businesses in society, such as car testing or dental appointments. It is inexpensive, saves the environment and there are studies that suggest it is more effective than sending physical letters. In this study, we intend to investigate whether SMS reminders, electronic letters, and physical letters for screening lead to increased participation and thus to a higher proportion of detected, treatable precursors of cervical cancer compared to before.

DETAILED DESCRIPTION:
Non-participation in the cervical screening program and sub-optimal follow-up after abnormalities or infection with a highly oncogenic HPV type detected in screening are the main risk factors for cervical cancer. Given this, It is important to reduce barriers to screening and facilitate participation in the screening program of cervical cancer. Offering self-sampling kits for human papillomavirus (HPV) testing has been examined in several research studies as a way to reach women who have not responded to screening invitations. Women who have been lost to follow-up can also be reached with self-sampling.

The purpose of this study is to investigate whether SMS reminders and electronic letters for screening attendance will increase participation compared to the current method where reminders are sent out with physical letters. In this study, women a with high risk of developing cervical cancer, due to not fully participating in screening or being followed up optimally, will be invited. Women are identified through registry linkages annually that examine screening history and status using a risk algorithm. Women receive an SMS or an electronic letter with an offer to request a self-sampling kit via the internet. Women with a higher risk for cervical cancer can be offered a self-sampling kit sent directly to their home address. The self-sampling kit comes with an instruction on how to take the sample and a postage-free answer envelope.

Submitted samples are analyzed with an approved and accredited method (Cobas 4800, Roche) that analyzes for HPV 16, HPV18 and other oncogenic HPV types. As the screening program changed the accredited HPV test in 2022 (to BD Onclarity), that test will be used from the timepoint of the change and onwards.

In the pilot of the study, follow-up is defined as follows:

1. For those women who are at the highest risk (previous glandular cell changes without follow-up), all HPV-positive women are referred via SMS directly to a women's clinic for investigation. HPV-negative women in this group have no increased risk and receive a text message with a calming message.
2. Women of an age above the screening program but who have either had a cell change that is not followed up or who have not participated at all in the last 10 years are treated in the same way as in paragraph 1.
3. Finally, the women of screening age who have not taken a cell sample for more than 15 years are identified. This group receive an SMS and HPV-positive women are referred, via SMS, for renewed sampling by a specially trained so-called dysplasia midwife. The sample is now being analyzed for both cytology and HPV. If the woman is HPV positive in both tests and in the case of deviating cytology, the woman is referred to a women's clinic. In other cases a text message with a reassuring message is sent.

The study has the usual level of confidence (p <0.05 two-sided) and statistical power (80%) the ability to demonstrate an increase of participation by 3 times or more.

The protocol was piloted in the Region of Skåne in 2019 and then rolled out nationally in 2020.

The study is rolled out nationally with annual linkages to identify women with an excess risk for cervical cancer and an adaptive approach to reaching women with SMS, electronic letters, and physically letters with direct delivery of HPV self-sampling kits or an option to order a self-sampling kid (depending on risk). The study is coordinated centrally and each region has a contact person to whom women who need follow-up are referred.

ELIGIBILITY:
Inclusion Criteria:

* Women resident in Region Skane who either: 1) have had glandular cell transformation that has not been followed-up, 2) are older than 65 years and have had cell transformation that has not been followed-up or who have not participated in screening during the last 10 years, 3) women who have not been screened for more than 15 years.

Exclusion Criteria:

* No exclusion except those who do not consent.

Ages: 33 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only women have a cervix
Enrollment: 20000 (Estimated)
Dates: Start 2019-08-19 (Actual); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of women responding to summon | Measured from the date of the summons until 12 months after the summons
  Participation rate in screening after summons.

SECONDARY OUTCOMES:
Number of positive screens | Measured from the date of the summons until 12 months after the summons
  Screening test results
Rate of precursors of cancer | Measured from the date of the summons until 12 months after the summons
  Cytologically and histopathologically confirmed percursors of cervical cancer.
Rate of cancer | Measured from the date of the summons until 12 months after the summons
  Histopathologically confirmed cervical cancers.

CONTACTS AND LOCATIONS:
Overall Officials: Miriam Elfström, PhD, Principal Investigator — Karolinska Institutet
Locations (6):
- Sweden (6):
  - Northern Region, Luleå, Norrbotten County
  - Southern Region, Lund, Skåne County
  - Western Region, Gothenburg, Västra Götaland County
  - Southeast Region, Jönköping
  - Region of Stockholm-Gotland, Stockholm
  - Region of Middle Sweden, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elfstrom KM, Sundstrom K, Andersson S, Bzhalava Z, Carlsten Thor A, Gzoul Z, Ohman D, Lamin H, Eklund C, Dillner J, Tornberg S. Increasing participation in cervical screening by targeting long-term nonattenders: Randomized health services study. Int J Cancer. 2019 Dec 1;145(11):3033-3039. doi: 10.1002/ijc.32374. Epub 2019 May 10. PMID 31032904
- [Result] Arroyo Muhr LS, Wang J, Hassan SS, Yilmaz E, Elfstrom MK, Dillner J. Nationwide registry-based trial of risk-stratified cervical screening. Int J Cancer. 2025 Jan 15;156(2):379-388. doi: 10.1002/ijc.35142. Epub 2024 Aug 15. PMID 39146489
- [Result] Wang J, Elfstrom KM, Borgfeldt C, Dillner J. A pilot study of risk-stratified cervical cancer screening. Open Res Eur. 2022 Sep 1;1:84. doi: 10.12688/openreseurope.13398.2. eCollection 2021. PMID 37645164